CLINICAL TRIAL: NCT03659591
Title: Triple Aim Psychotherapy: an RCT Comparing Cognitive Behaviour Therapy (CBT) to Adaptive Psychological Training (APT) - a Treatment Aimed at Improving Patient Experience, Population Health, and Cost-effectiveness
Brief Title: Triple Aim Psychotherapy: Aimed at Improving Patient Experience, Population Health, and Cost
Acronym: TAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Joseph Brant Hospital (Other)
Responsible Party: Principal Investigator, Dr. Steven Selchen, Chief of Psychiatry, Joseph Brant Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000-044-18
Record Dates: First submitted 2018-08-30; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Anxiety Symptoms; Depressive Symptoms
Keywords: Cognitive Behaviour Therapy; Community Mental Health; Adaptive Psychological Training; Quality of Life; Wellbeing; Treatment
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy; APT

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behaviour Therapy (Active Comparator): 10 week, manual-based group CBT treatment for depression and anxiety, followed by optional booster sessions
  Interventions: Behavioral: Cognitive Behaviour Therapy
- Adaptive Psychological Training (Active Comparator): 5 week, manual-based group APT treatment for depression and anxiety, followed by optional booster sessions
  Interventions: Behavioral: Adaptive Psychological Training

INTERVENTIONS:
Behavioral: Cognitive Behaviour Therapy — CBT will be delivered in group format, consisting of 10 weekly two-hour sessions, with 10 participants per group
  Other Names: CBT
  Arms: Cognitive Behaviour Therapy
Behavioral: Adaptive Psychological Training — APT will be delivered in group format, consisting of 5 weekly two-hour sessions, with 20 participants per group
  Other Names: APT
  Arms: Adaptive Psychological Training

SUMMARY:
Community mental health programs in publically-funded jurisdictions such as Canada often have limited budgets in order to provide services, which can result in inadequate access to effective treatment for patients. Cognitive Behaviour Therapy (CBT) is a gold-standard psychotherapy for depression and anxiety. In order to improve access to treatment, community mental healthcare settings often provide CBT in a group format for patients experiencing mild-to-moderate symptoms. However, typical protocols for delivering group CBT in a community setting nonetheless require a considerable investment of limited clinician time. The Institute for Healthcare Improvement (IHI) developed the Triple Aim, which is a framework describing an approach to optimizing health system performance by simultaneously pursuing three dimensions, namely improving the patient experience of care; improving the health of populations; and reducing the associated per capita costs of care. Adaptive Psychological Training (APT) is a group-based psychotherapy designed with all of the dimensions of the Triple Aim in mind simultaneously. In its development, APT drew heavily upon mindfulness-based approaches. To-date, APT has already demonstrated positive outcomes in pilot research and in community clinical settings. The purpose of the current study is to determine whether for a given population of patients experiencing mild-to-moderate symptoms of depression and/or anxiety, APT can facilitate meaningful change for more patients per time spent by clinicians than can CBT.

DETAILED DESCRIPTION:
Depression and anxiety are highly prevalent in the general population. Community mental health programs in publically-funded jurisdictions such as Canada often have relatively limited, fixed budgets in order to provide services, which can result in inadequate access to effective treatment for patients. Cognitive Behaviour Therapy (CBT) is a gold-standard psychotherapeutic treatment for depression and anxiety. In order to improve access to treatment, community mental healthcare settings often provide CBT in a group format for patients experiencing mild-to-moderate symptoms. However, typical protocols for delivering group CBT in a community setting nonetheless require a considerable investment of limited clinician time.

The question arises as to whether this is the most efficient and effective use of clinician time; in other words, per hour spent of clinician time, does this approach maximize the number of patients experiencing adequate and meaningful clinical improvement? The Institute for Healthcare Improvement (IHI) developed the Triple Aim, which is a framework describing an approach to optimizing health system performance by simultaneously pursuing three dimensions, namely improving the patient experience of care; improving the health of populations; and reducing the associated per capita costs of care. Studies of psychotherapy rarely pursue all three of these dimensions simultaneously. Efforts to achieve the best clinical outcome for an individual often lead to restrictive inclusionary/exclusionary criteria that sacrifice reaching the wider population; conversely, efforts to improve population health often prioritize composite overall clinical improvement across an entire group, even though the change experienced by many of the individuals in the population might not be clinically meaningful; focusing primarily on cost-effectiveness often sacrifices the individual's experience and/or the population's needs.

Adaptive Psychological Training (APT) is a group-based psychotherapy designed with all of the dimensions of the Triple Aim in mind simultaneously. In its development, APT drew heavily upon Mindfulness-Based Cognitive Therapy, an evidence-based psychotherapy that itself draws upon both evidence-based eastern psychotherapeutic practices and CBT, but APT also drew upon other evidence-based and evidence-supported psychotherapies including interpersonal and relational approaches, as well as meaning-focused psychoanalytic models. It also drew from psychology and neuroscience more broadly, as well as from learning theory and from practical clinical and operational experience. Inclusion/exclusion criteria, group size, number of sessions, in-session practice and learning, and between-session practice and learning were all adapted from the perspective of trying to achieve high quality outcomes for a broader population within more contained costs, and thereby increase access to quality care.

To-date, APT has already demonstrated positive outcomes in pilot research and in community clinical settings. The purpose of this specific study is to determine whether for a given population of patients experiencing mild-to-moderate symptoms of depression and/or anxiety, APT can facilitate meaningful change for more patients per time spent by clinicians than can CBT (the gold standard). The significance of this study includes its potential contribution to determining how best to deploy the limited resource of clinician time in a community setting in order to best help the most people.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-seeking adults, interested and willing to participate in group psychotherapy
* Mild-to-moderate depressive (score of ≥10 and <20 on PHQ9) and/or anxious (score of ≥8 and <15 on GAD7) symptoms
* Ability to communicate, in written and spoken English

Exclusion Criteria:

* Severe depressive/anxious symptoms
* Patients where the primary clinical focus is active suicidality or harm-to-others, psychosis, mania, substance use, posttraumatic stress, or personality pathology such that it would interfere with group function
* Recent course(s) of the study psychotherapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Triple Aim Measure | At 10 weeks; in a secondary fashion, this outcome will also be examined every two weeks across 6 months
  Numerator: The number of patients achieving reliable recovery; denominator: clinician time spent in hours ('reliable recovery' is defined as scores below 'caseness' for both depression [<10 on Patient Health Questionnaire (PHQ-9)] and anxiety [<8 on Generalized Anxiety Disorder-7 (GAD-7)], with any change from above caseness to below caseness meeting the threshold of the Reliable Change Index)

SECONDARY OUTCOMES:
Triple Aim Measure - recovery only | At 10 weeks; in a secondary fashion, this outcome will also be examined every two weeks across 6 months
  Triple Aim Composite Score (as above), but without the Reliable Change Index requirement
Triple Aim Measure - improvement only | At 10 weeks; in a secondary fashion, this outcome will also be examined every two weeks across 6 months
  Triple Aim Composite Score (as above), but without the remission requirement
Change from baseline - depressive symptoms | Pre- (week 0) and repeated every two weeks across 6 months
  Scale used to measure depressive symptoms is the Patient Health Questionnaire (PHQ-9); score ranges from 0-27, where higher values indicate more depressive symptoms (worse outcome)
Change from baseline - anxiety symptoms | Pre- (week 0) and repeated every two weeks across 6 months
  Scale used to measure anxiety symptoms is the Generalized Anxiety Disorder 7-item (GAD-7) Scale; score ranges from 0-21, where higher values indicate more anxiety symptoms (worse outcome)
Change from baseline - function | Pre- (week 0) and repeated monthly across 6 months
  Scale used to measure function is the World Health Organization Disability Assessment Schedule 2.0 - 12 item version (WHODAS 2.0 12-item); score ranges from 0-48, where higher values indicate lower functioning (worse outcome)
Change from baseline - mental wellbeing | Pre- (week 0) and repeated monthly across 6 months
  Scale used to measure mental wellbeing is the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS); score ranges from 14-70, where higher values indicate greater mental wellbeing (better outcome)
Change from baseline - self-compassion | Pre- (week 0) and repeated monthly across 6 months
  Scale used to measure self-compassion is the Self-Compassion Scale - Short Form (SCS-SF); score ranges from 12-60, where higher values indicate greater self-compassion (better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Selchen, MD MSt FRCPC, Principal Investigator — Joseph Brant Hospital
Locations (1):
- Joseph Brant Hospital, Burlington, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No